CLINICAL TRIAL: NCT06144268
Title: Evaluation of Live Birth Rate After Sperm Selection Using Microfluidic Technology (ZyMōt Multi (850µL) Sperm Separation Device) for Intra Uterine Insemination.
Brief Title: Live Birth Rate After Sperm Selection Using ZyMōt Multi (850µL) Device for Intra Uterine Insemination
Acronym: FERTINSEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC-2023-257
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-10

CONDITIONS: Infertility; Fertility Disorders
Keywords: Intra Uterine Insemination; Live birth; Microfluidic sperm selection
MeSH Terms: conditions — Infertility | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Density Gradient Centrifugation (DGC) (Active Comparator): During this procedure, raw semen sample is placed on 2 gradients: a lower phase (80%) and an upper phase (40%) followed by centrifugation. The composition of the gradients include a colloidal suspension of silica particles. At the end of centrifugation, each spermatozoa is situated at the gradient level that matches its density. The highly motile, morphologically normal, viable spermatozoa form a pellet at the bottom of the tube.
  Interventions: Other: Density Gradient Centrifugation
- ZyMōt Multi (850µL) (Experimental): ZyMōt Multi (850µL) is a flow-free dual chambered single-use device. The first chamber contains a sample inlet and a fluid channel separated from the second collection chamber by an 8-μm microporous membrane. Channel dimension and membrane porosity are designed to optimize the sorting and collection of the most motile sperm. Sorting is accomplished by the passage of sperm through the micropores of the membrane. This procedure does not require any preliminary semen processing, all centrifugation steps being eliminated.
  Interventions: Device: ZyMōt Multi (850µL)

INTERVENTIONS:
Device: ZyMōt Multi (850µL) — An amount of 850 µl untreated semen sample will be loaded into the inlet chamber with a help of a sterile insulin-type syringe. A volume of 750 µl of Sage Quinn's AdvantageTM Medium with Hepes + 5% HSA-solution medium will be placed on top of the membrane (outlet chamber). After 30 min of incubation in a humidified incubator (37°C), 500 µl of medium, containing the selected spermatozoa, will be retrieved from the upper side of the membrane (retrieval chamber). An amount of 400 µl will be necessary for the IUI procedure.
  Other Names: FERTILE Plus® device (KOEK EU GmbH, Biotechnology)
  Arms: ZyMōt Multi (850µL)
Other: Density Gradient Centrifugation — The gradient columns will be prepared by placing 1 ml 80% gradient media in a centrifuge tube and an additional 1 ml of 40% gradient layered on top.
  The raw semen sample will be placed on top of the gradient (1ml semen/gradient tube) and centrifuged at 300xg for 20 minutes. The sperm pellet will be collected and washed 2 times for 5 min at 800xg in Sage Quinn's AdvantageTM Medium with Hepes + 5% HSA-solution.
  The resulted pellet will be resuspended in the washing solution in a volume that will provide at least 1x106 forward motile spermatozoa in 400 µl, as this amount is necessary for IUI procedure.
  Arms: Density Gradient Centrifugation (DGC)

SUMMARY:
This single centre interventional pilot randomized control study intends to compare two methods of sperm preparation for couples referred for Intra Uterine Insemination (IUI) procedure. Couples will be randomly allocated to one of the two sperm selection methods: Density Gradient Centrifugation (DGC, standard) or ZyMōt Multi (850µL) device (treatment) groups. The study will compare the live birth rate (number of live births per number of IUI procedures) between the treatment and standard groups.

DETAILED DESCRIPTION:
Intrauterine insemination is a commonly used method for Medically Assisted Reproduction for patients with mild male factor infertility, anovulation, endometriosis, and unexplained infertility. It is also the procedure of choice in cases of lesbian couples or single women, using donor sperm.

During the IUI procedure, the sperm suspension is introduced into the uterus through the cervix canal using an insemination catheter containing 0.4 ml sperm. Before sperm can be used in IUI, it must first be processed. The aim of semen preparation is to select the best sperm cell population (highly motile, morphologically normal spermatozoa with minimal DNA damage) with the highest fertilization potential.

One of the most used sperm preparation technique is DGC. This technique allows the separation of sperm cells based on their density. Morphologically normal and abnormal spermatozoa have different densities. A mature morphologically normal spermatozoon has a slightly higher density, whereas an immature and morphologically abnormal spermatozoon has a lower density. During this procedure, raw semen sample is placed on 2 gradients: a lower phase (80%) and an upper phase (40%) followed by centrifugation. The composition of the gradients include a colloidal suspension of silica particles. At the end of centrifugation, each spermatozoa is situated at the gradient level that matches its density. The highly motile, morphologically normal, viable spermatozoa form a pellet at the bottom of the tube. This procedure is relatively easy to perform but both the centrifugation steps and the silica particle are considered to have a negative impact on DNA integrity.

Recently, microfluidic technology was introduced as an alternative to the conventional sperm sorting techniques. As this procedure does not require semen processing, it reduces the sperm preparation time and eliminates sperm DNA damaging procedures (e.g. by centrifugation). This technology is a chemical-free method of sorting healthy normal sperm using a sterile disposable ZyMōt Multi (850µL) sperm separation device. Sperm selected by this device proved to have better motility and less DNA damage compared to DGC procedure. More recently, the efficacy of this device has been reported to significantly increase ongoing pregnancy rate when compared with DGC in IUI cycles. However, large, correct studies that investigate live birth rate are missing.

The present study aims to determine whether the use of ZyMōt Multi (850µL) device for sperm selection improves the live birth rate in IUI patients as compared to the standard DGC procedure. Couples undergoing IUI procedure will be included in the study if they are planned for IUI with fresh autologous ejaculate.

Patients that fulfill the inclusion criteria will be randomly allocated to one of the two sperm selection methods: DGC (standard) or ZyMōt Multi (850µL) device (treatment) groups. The randomization will be performed based on an electronically generated list. A patient participation to the study will be limited to 3 consecutive IUI attempts (within a period of 6 months). Same semen preparation protocol used in the 1st IUI attempt [ZyMōt Multi (850µL) or DGC] will be used in the next 2 consecutive IUIs. Following the IUI procedure (with sperm selected with either one of the two methods), the patients will be monitored for pregnancy, clinical pregnancy and neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Fresh autologous ejaculate
* Female age: <37 at start of the first insemination
* 1st IUI ever here, maximum 3 consecutive IUIs during max 6 months
* BMI <35
* All natural cycles, ovulation induction allowed
* Presence of 1 or 2 follicles at the last ultrasound
* Regular menses (26-35 days)
* >1 million Total Progressive Motile Sperm Count (TPMC) after previous routine capacitation with DGC
* Presence of at least 1 potent tube after Hyfosy

Exclusion Criteria:

* Presence of intracavitary pathology at ultrasound
* Evidence of advance endometriosis (Grade 3 and 4)

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate after 3 consecutive IUIs | 9 months following IUI
  Number of live births per number of inseminations

SECONDARY OUTCOMES:
Pregnancy rate | 14 days following IUI
  number of pregnancies (positive hCG) per number of inseminations
Miscarriages rate | 12 weeks following IUI
  number of miscarriages per number of inseminations

CONTACTS AND LOCATIONS:
Overall Officials: Shari Mackens, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel CRG, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
The results of the study will be publicly disseminated following submission in peer-reviewed scientific journals.

REFERENCES:
- [Result] Gode F, Bodur T, Gunturkun F, Gurbuz AS, Tamer B, Pala I, Isik AZ. Comparison of microfluid sperm sorting chip and density gradient methods for use in intrauterine insemination cycles. Fertil Steril. 2019 Nov;112(5):842-848.e1. doi: 10.1016/j.fertnstert.2019.06.037. Epub 2019 Sep 19. PMID 31543253